CLINICAL TRIAL: NCT01147783
Title: A Comparison of Pediatric Airway Anatomy With the SimBaby High-Fidelity Simulator
Brief Title: Airway Anatomy of the SimBaby
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Oliver Kimberger, M.D., P.D., Medical University of Vienna, Dept. of Anesthesia, Genereal Intensive Care and Pain Management
Other Study IDs: Anae-Vie-SimbabyCT
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-06

CONDITIONS: Airway Reality
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SimBaby
  Interventions: Other: CT, MRI
- Infants (1-12 mo)
  Interventions: Other: CT, MRI

INTERVENTIONS:
Other: CT, MRI

SUMMARY:
The aim of the present study is to compare radiographic upper airway measurements of the SimBabyTM pediatric patient high-fidelity simulator with actual human airway anatomy to assess the grade of realism of the simulator.

ELIGIBILITY:
Inclusion Criteria:

* MRI or CT head or neck including upper airway
* age: 1-12 months

Exclusion Criteria:

* no pathology of airway, face, neck
* no airway device in place
* head not in neutral position
* neck collar

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants undergoing routine head MRI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
pharyngeal measurements

SECONDARY OUTCOMES:
anatomic structures of the upper airway
  distances, volumes and cross sectional areas of the tongue, soft palat, pharyngeal structures as well as oral airspace

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, M.D., P.D., Principal Investigator — Medical University of Vienna, Dept. of. Anesthesia, General Intensive Care and Pain Management
Locations (1):
- Medical University of vienna, Vienna, Austria

REFERENCES:
- [Derived] Schebesta K, Hupfl M, Ringl H, Machata AM, Chiari A, Kimberger O. A comparison of paediatric airway anatomy with the SimBaby high-fidelity patient simulator. Resuscitation. 2011 Apr;82(4):468-72. doi: 10.1016/j.resuscitation.2010.12.001. Epub 2011 Jan 14. PMID 21237552